CLINICAL TRIAL: NCT03012815
Title: A Prospective Randomized Controlled Open Label Trial of Symptom-triggered Benzodiazepine Versus Fixed-dose Gabapentin for Alcohol Withdrawal Syndrome
Brief Title: Gabapentin for Alcohol Withdrawal Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ruth E Bates, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-008712
Record Dates: First submitted 2016-12-27; First posted 2017-01-06 (Estimated); Results first posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Alcohol Withdrawal Syndrome
Keywords: gabapentin; Alcohol Withdrawal Syndrome; benzodiazepine; symptom-triggered
MeSH Terms: interventions — Gabapentin; Benzodiazepines; Lorazepam; Chlordiazepoxide; Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gabapentin (Experimental): Patients will receive gabapentin taper over 9 days with the option to add divalproex for patients who have a history of seizures or severe withdrawal. Will still undergo CIWA-Ar scoring but will not be administered a benzodiazepine.
  Interventions: Drug: Gabapentin; Drug: Divalproex Sodium
- Benzodiazepine (Active Comparator): Patients will receive a benzodiazepine if scoring greater than 9 on the CIWA-Ar scale.
  Interventions: Drug: Benzodiazepines

INTERVENTIONS:
Drug: Gabapentin — Gabapentin administered as a taper
  Other Names: Neurontin
  Arms: Gabapentin
Drug: Benzodiazepines — Benzodiazepines administered using a symptoms triggered protocol
  Other Names: lorazepam; chlordiazepoxide
  Arms: Benzodiazepine
Drug: Divalproex Sodium — Given in addition to gabapentin in high risk patients (i.e. seizures, TBI history, DT history)
  Other Names: Depakote
  Arms: Gabapentin

SUMMARY:
The current "gold-standard" for the management of alcohol withdrawal syndrome (AWS) is symptom-triggered administration of benzodiazepines. This method of treatment has several drawbacks that have been described in the literature. Thus benzodiazepine sparing agents have been evaluated for use in AWS. One of these agents that has not only shown benefit for AWS but also benefits on complete abstinence, reducing a return to heavy drinking, and cravings is gabapentin. In clinical practice at Mayo Clinic gabapentin is used for this purpose. Due to the limited reports of the safety and efficacy of a protocol involving gabapentin for AWS, a study to compare gabapentin to symptom-triggered lorazepam will be completed.

DETAILED DESCRIPTION:
The current "gold-standard" for the management of alcohol withdrawal syndrome is symptom-triggered administration of benzodiazepines. Benzodiazepines and use of a symptom-triggered approach has several drawbacks such as over administration of medication due to many subjective patient reported symptoms. Benzodiazepines may contribute to a drug-induced delirium or high dosage may necessitate transfer to an ICU setting. Abrupt withdrawal of benzodiazepines also contribute to cravings, rebound insomnia, and anxiety that have been shown to increase the risk of a return drinking.

Clinical use of gabapentin for alcohol withdrawal has been presented by Maldonado at Stanford University Hospitals. (Academy of Psychosomatic Medicine Annual Meeting, 2013-2015) At Mayo Clinic, the Psychiatry Consultation-Liaison hospital service has been recommending the use of a modified gabapentin protocol since January 2015, which has been clinically accepted on medical, surgical, and psychiatric hospital services. The purpose of this research is to investigate the reactive benzodiazepine versus proactive gabapentin approaches to AWS in a prospective, randomized, open-label study.

ELIGIBILITY:
Inclusion criteria

1. Prediction of Alcohol Withdrawal Severity Scale (PAWSS) score >4.
2. Adults age 18 or older.
3. Sufficient understanding of English.
4. Hospitalized on Hospital Internal Medicine or Generose.

Exclusion criteria

1. Severe renal impairment (estimated CrCl < 30).
2. Intensive Care Unit (ICU) level of care.
3. Not responsive due to alcohol intoxication or withdrawal.
4. Already taking gabapentin more than 300 mg three times a day.
5. Prescribed pregabalin.
6. Primary seizure disorder.
7. Acute benzodiazepine withdrawal.
8. Concurrent substance use disorders (such as opioid use disorder, stimulant use disorder) if the disorder is assessed to be clinically significant. Cannabis use disorder will be allowed.
9. Concurrent anticonvulsant medications for psychiatric indications (e.g. bipolar disorder) will be allowed.
10. Pregnancy.
11. Involuntary legal status (e.g., on court commitment).
12. Patients admitted greater than 12 hours prior to potential enrollment.
13. Patients receiving therapeutic dose of gabapentin (rather than continuation of home dose) prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth E Bates, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Furieri FA, Nakamura-Palacios EM. Gabapentin reduces alcohol consumption and craving: a randomized, double-blind, placebo-controlled trial. J Clin Psychiatry. 2007 Nov;68(11):1691-700. doi: 10.4088/jcp.v68n1108. PMID 18052562
- [Background] Leung JG, Hall-Flavin D, Nelson S, Schmidt KA, Schak KM. The role of gabapentin in the management of alcohol withdrawal and dependence. Ann Pharmacother. 2015 Aug;49(8):897-906. doi: 10.1177/1060028015585849. Epub 2015 May 12. PMID 25969570
- [Background] Maldonado JR, Sher Y, Das S, Hills-Evans K, Frenklach A, Lolak S, Talley R, Neri E. Prospective Validation Study of the Prediction of Alcohol Withdrawal Severity Scale (PAWSS) in Medically Ill Inpatients: A New Scale for the Prediction of Complicated Alcohol Withdrawal Syndrome. Alcohol Alcohol. 2015 Sep;50(5):509-18. doi: 10.1093/alcalc/agv043. Epub 2015 May 21. PMID 25999438
- [Derived] DeFoster RE, Morgan RJ 3rd, Leung JG, Schenzel H, Vijapura P, Kashiwagi DT, Fischer KM, Philbrick KL, Kung S. Use of Gabapentin for Alcohol Withdrawal Syndrome in the Hospital Setting: A Randomized Open-Label Controlled Trial. Subst Use Misuse. 2023;58(13):1643-1650. doi: 10.1080/10826084.2023.2236223. Epub 2023 Jul 19. PMID 37469099
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Gabapentin: Patients received gabapentin taper over 9 days with the option to add divalproex for patients who have a history of seizures or severe withdrawal. Still underwent CIWA-Ar scoring but did not receive a benzodiazepine.
  Gabapentin: Gabapentin administered as a taper
  Divalproex Sodium: Given in addition to gabapentin in high risk patients (i.e. seizures, TBI history, DT history)
- Benzodiazepine: Patients received a benzodiazepine if scoring greater than 9 on the CIWA-Ar scale.
  Benzodiazepines: Benzodiazepines administered using a symptoms triggered protocol
Period: Overall Study
Arm/Group | Gabapentin | Benzodiazepine
Started | 46 | 42
Completed | 41 | 40
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 3 | 2
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Benzodiazepine | Total
Number analyzed (Participants) | 46 | 42 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (13.51) | 46.7 (11.88) | 47.6 (12.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 23
  Male | 32 | 33 | 65
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 46 | 42 | 88

OUTCOME MEASURES:

1. Primary Outcome: Mean Length of Hospital Stay
Description: The length of hospital stay for Alcohol withdrawal syndrome. The time interval between admission and either discharge or the time at which Clinical Institute Withdrawal Assessment - Alcohol revised (CIWA-Ar) scores are <10 for 36 hours (up to 240 hours). Measured in hours. CIWA-Ar measures severity of 10 observed or measured alcohol withdrawal signs or symptoms. Zero to 7 points are assigned to each item, except for the last item, which is assigned 0-4 points, with a total possible score of 67. Total score ranges from 0 (best possible outcome)-67 (worst possible outcome). Lower scores (0-8) represent fewer withdrawal symptoms and less severity, scores > 8 represent more withdrawal symptoms and greater severity
Time Frame: Time to discharge or time to CIWA-Ar score < 10 for 36 hours (whichever came first) up to 240 hrs.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Gabapentin | Benzodiazepine
Number analyzed (Participants) | 46 | 42
hours | 44.91 (12.17) | 50.50 (25.07)

2. Secondary Outcome: Number of Participants With Delirium Tremens (DT)
Description: The number of participants experiencing delirium tremens during their hospitalization (between admission and discharge).
Time Frame: During hospitalization (up to 240 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin | Benzodiazepine
Number analyzed (Participants) | 46 | 42
Participants | 0 | 0

3. Secondary Outcome: Maximun Alcohol Withdrawal Severity Per CIWA-Ar Scale
Description: CIWA-Ar measures severity of 10 observed or measured alcohol withdrawal signs or symptoms. Zero to 7 points are assigned to each item, except for the last item, which is assigned 0-4 points, with a total possible score of 67. Total score ranges from 0 (best possible outcome)-67 (worst possible outcome). Lower scores (0-8) represent fewer withdrawal symptoms and less severity, scores > 8 represent more withdrawal symptoms and greater severity
Time Frame: 4 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gabapentin | Benzodiazepine
Number analyzed (Participants) | 46 | 42
score on a scale | 13.15 (5.70) | 12.81 (6.94)

4. Secondary Outcome: Change in Sleepiness as Assessed by the Epworth Sleepiness Scale
Description: The ESS is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. Most people engage in those activities at least occasionally, although not necessarily every day. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP), or their daytime sleepiness.
Time Frame: Baseline and 2 days
Population: Those patients who completed baseline questionnaire and follow-up questionnaire 48 hours later
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gabapentin | Benzodiazepine
Number analyzed (Participants) | 19 | 10
score on a scale | -0.03 (4.02) | 0.07 (5.35)

5. Secondary Outcome: Mean Total Benzodiazepine Use
Description: The total amount of benzodiazepines administered. Measured by lorazepam equivalent, mg.
Time Frame: Time to discharge or time to CIWA-Ar score < 10 for 36 hours (whichever came first) up to 240 hrs.
Measure: Mean (Standard Deviation); unit: milligrams
Groups:
- Gabapentin: Patients received gabapentin taper over 9 days with the option to add divalproex for patients who have a history of seizures or severe withdrawal.
  Gabapentin: Gabapentin administered as a taper
  Divalproex Sodium: Given in addition to gabapentin in high risk patients (i.e. seizures, TBI history, DT history)
Arm/Group | Gabapentin | Benzodiazepine
Number analyzed (Participants) | 46 | 42
milligrams | 5.2 (6.8) | 10.8 (14.9)

6. Secondary Outcome: Number of Participants Experiencing Seizure
Description: The number of subjects who developed seizure during their hospitalization.
Time Frame: During hospitalization (up to 240 hours).
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin | Benzodiazepine
Number analyzed (Participants) | 46 | 42
Participants | 0 | 0

7. Secondary Outcome: Change in Cravings as Assessed by the Penn Alcohol Craving (PACS) Scale
Description: PACS is a 5 item self-rated scale of alcohol craving (0 = none to 6 = strong urge). Total scores range from 0 (little craving for alcohol) to 30 (irresistible urge to drink alcohol)
Time Frame: Baseline and 2 days
Population: Those patients who completed baseline questionnaire and follow-up questionnaire 48 hours later
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gabapentin | Benzodiazepine
Number analyzed (Participants) | 19 | 10
score on a scale | -8.12 (9.15) | -8.45 (7.89)

8. Secondary Outcome: Change in Anxiety Symptoms as Measured by the Generalized Anxiety Disorder-7 (GAD-7) Scale
Description: GAD-7 is GAD-7 is a 7-item self-administered scale of Generalized Anxiety Disorder symptoms (0 = not at all to 3 = nearly every day). Total scores range from 0 to 21. Total scores of 0-4 = minimal anxiety, Total scores of 5-9 = mild anxiety, total scores of 10-14 = moderate anxiety and total scores of 15-21 = severe anxiety.
Time Frame: Baseline and 2 days
Population: Those patients who completed baseline questionnaire and follow-up questionnaire 48 hours later
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gabapentin | Benzodiazepine
Number analyzed (Participants) | 19 | 10
score on a scale | -0.07 (4.80) | -3.79 (6.08)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the patient's hospitalization (from admission to discharge, up to 240 hours).
Arm/Group | Gabapentin | Benzodiazepine
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/42
Serious Adverse Events (participants affected / at risk) | 1/46 | 0/42
Other Adverse Events (participants affected / at risk) | 0/46 | 0/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin (N=46) | Benzodiazepine (N=42)
Allergic reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Angioedema attributed to allergic reaction to gabapentin

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/15/NCT03012815/Prot_SAP_000.pdf